CLINICAL TRIAL: NCT01095939
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Benazepril (ATC N° C09AA07) in the Treatment of Persistent Renal Dysfunction in Pre-eclamptic Women
Brief Title: Post-preeclampsia Renal Project: Study of Nephroprotection in Women Having Suffered Preeclampsia
Acronym: RPPEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Antoinette Pechere-Bertschi, MD, Dr, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-136
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Renal Alteration
Keywords: Renal function consecutive to pre-eclampsia
MeSH Terms: interventions — benazepril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Placebo Comparator)
  Interventions: Drug: Placebo
- Benazepril (Experimental)
  Interventions: Drug: Benazepril hydrochloride

INTERVENTIONS:
Drug: Placebo — Tablets; oral administration; once a day for 6 months. After this period of 6 months blinded treatment, the treatment will be stopped for 2 weeks. At the end of this washout period, a new renal evaluation is done. At that time, opened label treatment will be proposed to the women who still show renal alterations after a 2 weeks washout period
  Arms: Control Arm
Drug: Benazepril hydrochloride — Tablets (10 or 20 mg); oral administration; once a day for 6 months. After this period of 6 months blinded treatment, the treatment will be stopped for 2 weeks. At the end of this washout period, a new renal evaluation is done. At that time, opened label treatment will be proposed to the women who still show renal alterations after a 2 weeks washout period
  Other Names: Cibacen; Lotensin; ATC: C09AA07
  Arms: Benazepril

SUMMARY:
The purpose of the Post-preeclampsia Renal Project is to investigate the renal function of preeclamptic women after delivery, and to determine whether the anti-hypertensive drug named benazepril efficiently improves the dysfunctions observed.

DETAILED DESCRIPTION:
Several epidemiological studies suggest that the risk of death from cardiovascular causes among women with preeclampsia may be increased, and that preeclampsia contrary to what has been long thought, is not cured with delivery. Preeclampsia has long been considered a 2-stage disease, stage one corresponding to an impaired placental perfusion resulting from abnormal spiral artery remodeling, and stage two corresponding to the maternal manifestations of disease, characterized by hypertension and proteinuria. However, preeclampsia might include an additional, 3rd stage, that of the post-partum period (Gammill & Roberts, 2007) This phase deserves to be investigated. In particular, it is crucial to determine whether the changes that occur in renal hemodynamics during preeclampsia are reversible after more than 6 weeks, and whether PEC women are salt-sensitive after delivery.

The link between chronic kidney disease and cardiovascular mortality is well established. An independent, graded association exists between a reduced GFR and the risk of death, cardiovascular events, and hospitalization (Go et al, 2004). Besides, salt-sensitivity is associated with an increased cardiovascular and renal risk (Franco & Oparil, 2006). The Renal Post PEC study aims at establishing if the renal dysfunctions that occur in PEC women can be reversed by the administration of inhibitors of the renin-angiotensin system that are known to improve cardiovascular and renal risk profiles in hypertensive patients. By virtue of their potent renal vasodilatory properties and favourable remodelling of the GBM, ACE inhibitors may improve salt-sensitivity, endothelial function, renal plasma flow and GFR, and general renal prognosis in women who experienced from preeclampsia.

ELIGIBILITY:
Pre-selection Criteria:

* Normotensive women with no proteinuria before the 20th week of gestation AND
* Women with hypertension (BP ≥140/90 mm Hg) and proteinuria (≥ 0.3 g /24h or 2++ dipstick) after the 20th week of gestation

Inclusion Criteria:

* Clearance of creatinine ≤ 80 ml/min (Gault et Cockcroft)
* Serum creatinine ≥ 80 µmol/L
* Microalbuminuria comprised between 30 and 300 mg/d and/or a urinary spot with microalbuminuria/creatinine ratio ≥ 3.5 and/or macroalbuminuria (24h urinary albumin excretion ≥ 0.500 mg)
* BP ≥ 140/90 mm Hg OR ongoing antihypertensive treatment
* CRP ≥ 4 mg/dL

Exclusion Criteria:

* Those unlikely to co-operate in the study
* Those who refuse to use appropriate contraceptive measures during the treatment period (intrauterine device, oral contraceptives, condom, diaphragm)
* Those with a history of pre-term delivery
* Those with known history of severe allergic reaction
* Those who consume drugs
* Aged < 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
microalbuminuria excretion rate (spot or 24h) | Baseline; 1 week + 24 weeks after treatment start
eGFR | Baseline; 1 week + 24 weeks after treatment start

SECONDARY OUTCOMES:
Filtration fraction % | Baseline; 1 week + 24 weeks after treatment start
24h Ambulatory Blood Pressure | Baseline; 1 week and 24 weeks after treatment start
  Mean; diurnal; nocturnal
Effective Renal Plasma Flow | Baseline; 1 week and 48 weeks after treatment start
Adverse Events | From signature of informed consent until last follow-up visit (36 months after treatment start)

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Pechère, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Geneva University Hospitals, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne

REFERENCES:
- [Derived] Ditisheim A, Wuerzner G, Ponte B, Vial Y, Irion O, Burnier M, Boulvain M, Pechere-Bertschi A. Prevalence of Hypertensive Phenotypes After Preeclampsia: A Prospective Cohort Study. Hypertension. 2018 Jan;71(1):103-109. doi: 10.1161/HYPERTENSIONAHA.117.09799. Epub 2017 Nov 13. PMID 29133363